CLINICAL TRIAL: NCT04796051
Title: Comparison Between Effect of Posterior Cervical Weighting and Deep Cervical Flexion Exercise on Forward Head Posture: Randomized Control Trial
Brief Title: Comparison Between Effect of Posterior Cervical Weighting and Deep Cervical Flexion Exercise on Forward Head Posture
Acronym: FHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0305072
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2021-03

CONDITIONS: Postural Kyphosis; Neck Pain; Deformity of Spine; Deformity; Muscle Weakness; Neck Syndrome; Forward Head Posture; Brace
MeSH Terms: conditions — Neck Pain; Congenital Abnormalities; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: 61 healthy individuals aged 18-65 are planned to participate in our study. Each case will fill out a questionnaire and will be subjected to a detailed examination by checking whether there have any factors that would cause the participant to be excluded from the study. Participants meeting the criteria will be divided into two groups according to their degrees of craniovertebral angle (CVA) after their participation in the study is approved. Neck Injury Index: The scale consists of 20 questions, the intensity of the pain; researches in terms of recreational, professional, social and daily life functions and emotional factors. Each question consists of a 10 cm long visual analog scale. CVA above 52 degrees will be considered as normal head posture, while less than 48 degrees will be considered as forward head posture.
Who Masked: Outcomes Assessor
Masking Description: An external assessors would be invited to assess the study's participants before and after the treatment. The extensor assessor would be blind to which group he/she is assessing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck orthosis - posterior cervical weight (Experimental): The posterior cervical weight orthosis is made of a well-padded adjustable Velcro attached to the end with a two-kilogram weight attached with two durable straps. The device is firmly anchored around the curvature of the jaw and attached with Velcro to the apex of the skull. Neck orthosis group will use a cervical orthosis (with the posterior cervical neck weight) for 10 minutes / 3 times a day, for a total of 30 minutes a day
  Interventions: Device: Neck orthosis - with posterior cervical weight
- Deep cervical flexors exercise (Active Comparator): Deep cervical flexors exercise group will do 15 repetitions x 3 sets of deep neck flexor exercises every day of the week.
  Interventions: Other: Deep cervical flexors exercise

INTERVENTIONS:
Device: Neck orthosis - with posterior cervical weight — The posterior cervical weight orthosis is made of a well-padded adjustable Velcro attached to the end with a two-kilogram weight attached with two durable straps. The device is firmly anchored around the curvature of the jaw and attached with Velcro to the apex of the skull.
  Other Names: Posterior cervical neck weight - Azzkol Orthosis
  Arms: Neck orthosis - posterior cervical weight
Other: Deep cervical flexors exercise — The participant will lay down in crook lying position, participant's head relaxed on the flat surface. Each participant will passively tuck in his/her chin without activation of superficial cervical muscles. Participants of this group will do 15 repetitions x 3 sets of deep neck flexor exercises every day of the week.
  Other Names: Deep cervical flexors activation
  Arms: Deep cervical flexors exercise

SUMMARY:
It has been reported that the head protrudes forward relative to the body from the sagittal plane associated with the anterior shifting of the line of gravity (LOG) relative to the base of support (BOS). On the other hand, the center of gravity (COG) has changed with the forward head posture (FHP) and is related to mechanical and musculoskeletal modifications due to postural control, which affects the whole body balance. Griegel-Morris et al. Reported that, after evaluating eighty-eight healthy participants, 66% had a forward head posture (FHP). In addition, he stated that the inverted head posture in the forward head posture will not only cause neck problems, but also can extend to the shoulder joint and thoracic spine. As a result, it causes a general imbalance in the musculoskeletal system. Jung-Ho Kang and his colleagues examined the effect of daily sitting times of computer users on dynamic and static balance and stated that balance ability decreased in heavy computer users. Another study on forward head posture (IBP) revealed that it limits ankle joint movement, especially in ankle plantarflexion.

DETAILED DESCRIPTION:
One of the most common postural deformities in the neck region is forward head posture seen in 66% of the population according to the American Physical Therapy Association. The use of computers and smartphones and long readings, which are the result of today's technological lifestyle, is one of the most common causes of FHP, causing the body to lean forward for hours. Maintaining the reverse neck posture also forces the body into many bad postures that damage the spine. Although forward head posture is experienced unconsciously at first, this unbalanced posture will accompany various degrees of advanced head posture, which turns into deformity, symptoms and complications.

FHP is an anterior translation of the head characterized by the extension of the upper cervical vertebra C1 and 2 and the bending of the lower cervical vertebra. According to Kapandji, each inch (2.54 cm) of the head forward equals the extra 4.5 kg on the neck extensor muscle, which leads to muscle fatigue and weakness, resulting in an unbalanced head posture with an abnormal bow in the neck. Immunohistochemical studies conducted by Satoshi Inami and colleagues showed that there is damage to the synovial folds containing nociceptive nerve endings as a result of compression of the facet joints in the forward head posture.

Aim of the work The aim of this study is to present a neck orthosis to correct neck posture and to see how posture correction will reflect on balance and plantar pressure distribution in individuals with forward head posture. This study can help answer questions about changes in gait level and mechanics between the spine and peripheral levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over willing to attend the study.
* Individuals with craniovertebral angle (CVA) less than 48 degrees for those participating in forward head posture (FHP).
* Young adults without known problems will be divided into groups by evaluating their craniovertebral angle value. (As individuals below 48 degrees).
* Mechanical neck pain experienced / felt in the last 3 months.

Exclusion Criteria:

* Spine trauma, surgery, bone pathology, arthritis, etc. Having a history of illness.
* Kyphotic deformity types are rounded back, Scheuermann's disease, hunched back, flat back and Dowager hump.
* Any spinal deformity, bone abnormality, postural deformity, and disc herniation with / without peripheral symptoms.
* Body mass index (BMI)> 30, which is an indicator of obesity.
* Suffering from balance problems, coordination problems, and other neurological or vestibular diseases that affect body balance and posture.
* Any orthopedic or neurological disease affecting the body joints or the integrity of the musculoskeletal system.
* Use of any medication that can cause dizziness or drowsiness in the last months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Craniovertebral Angle (CVA) | 6 weeks
  Cranio vertebral angle: Above 52 degrees will be considered as normal head posture, while less than 48 degrees will be considered as forward head posture
Neck Disability Index (NDI) | 6 weeks
  The scale consists of 20 questions, the intensity of the pain; researches in terms of recreational, professional, social and daily life functions and emotional factors. Maximum score is 50 (which is total maximum score) means severe neck disability. Minimum score is 0(which is total minimum score) means without any reported neck disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ossama Ragai, PHD Prof, Principal Investigator — Alexandria University
Locations (1):
- Ethics Committee - Alexandria Faculty of Medicine, Alexandria, Egypt